CLINICAL TRIAL: NCT00720408
Title: A Randomized, Open-Label, Comparative, Multi-Center Study to Assess the Safety and Efficacy of Prograf (Tacrolimus)/MMF and Extended Release (XL) Tacrolimus /MMF and Steroid Withdraw in de Novo Liver Transplant Recipients.
Brief Title: A Randomized Study to Assess the Safety and Efficacy of Prograf vs Prograf-XL in de Novo Liver Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRGXLLTx-0702-TW
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Liver Transplantation; Transplantation Immunology; Host vs Graft Reaction
Keywords: Immunosuppressant; Graft loss; Combination drug therapy; Randomized controlled trial; Open level method
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf-XL + MMF (Experimental)
  Interventions: Drug: Prograf-XL; Drug: MMF
- Prograf + MMF (Active Comparator)
  Interventions: Drug: Prograf; Drug: MMF

INTERVENTIONS:
Drug: Prograf-XL — oral
  Other Names: tacrolimus extended release; FK506E; MR4
  Arms: Prograf-XL + MMF
Drug: Prograf — oral
  Other Names: tacrolimus; FK506
  Arms: Prograf + MMF
Drug: MMF — oral
  Other Names: Mycophenolate Mofetil

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Prograf extended release(XL) plus MMF with Prograf plus MMF and steroid withdrawal in de novo Liver transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures
* Patient is a primary liver transplant recipient
* Patient must receive first dose of XL or Prograf (or IV tacrolimus for subjects unable to tolerate oral study drug) within 48 hours of transplantation
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to transplant

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a liver
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Patient has received a liver transplant from a non-heart beating donor
* Patient has received an ABO incompatible donor liver
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except hepatocellular carcinoma within UCSF Criteria 21 and basal or non-metastatic squamous cell carcinoma of skin that has been treated successfully
* Patient has fulminant hepatic failure, unless hemodynamically stable
* Patient has an uncontrolled concomitant infection, a systemic infection requiring treatment (except viral hepatitis), or any other unstable medical condition that could interfere with the study objectives
* Patient has severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patient is currently taking or has been taking an investigational drug in the 30 days prior to transplant
* Patient has a known hypersensitivity to tacrolimus, mycophenolate mofetil or corticosteroids
* Patient is pregnant or lactating
* Patient is unlikely to comply with the visits scheduled in the protocol, including the protocol biopsies
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy confirmed acute rejection (local assessment of biopsies performed due to hepatic dysfunction) during the 6 months post-transplant. | 6 month

SECONDARY OUTCOMES:
Patient and graft survival rates during the 6 and 12 months post-transplant | 6 and 12 month
Incidence of biopsy confirmed acute rejection (local assessment of biopsies performed due to hepatic dysfunction) during the 12 months post-transplant | 12 month
Incidence of anti-lymphocyte antibody therapy for treatment of rejection during the 6 and 12 months post-transplant | 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (3):
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District